CLINICAL TRIAL: NCT01595984
Title: Randomized, Multicenter, Open-label, Comparative Study of Efficacy and Safety of Treatment With a Calcineurin Inhibitor (CNI), Associating Myfortic ® and Neoral ® Compared to a CNI-free Treatment, Combining Myfortic ® and Certican ® , in Adult Patients With de Novo Renal Transplant
Brief Title: Comparison of Efficacy and Safety of Treatment With a Calcineurin Inhibitor (CNI)Versus a CNI-free Treatment in Renal Transplantation (CIME)
Acronym: CIME
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI10-PR-CHOUKROUN; 2011-001385-18 (EudraCT Number)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Kidney Failure
Keywords: kidney; transplantation; graft; creatinin
MeSH Terms: conditions — Renal Insufficiency | interventions — Cyclosporine; Mycophenolic Acid; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporin + Mycophenolate mofetil (Active Comparator)
  Interventions: Drug: cyclosporin + mycophenolate mofetil
- Everolimus + mycophenolate mofetil (Experimental)
  Interventions: Drug: everolimus + mycophenolate mofetil

INTERVENTIONS:
Drug: cyclosporin + mycophenolate mofetil — antirejection drug, renal transplantation
  Arms: Cyclosporin + Mycophenolate mofetil
Drug: everolimus + mycophenolate mofetil — antirejection drug, renal transplantation
  Arms: Everolimus + mycophenolate mofetil

SUMMARY:
The main objective of this protocol is to compare the impact on renal function of two different immunosuppressive regimens in patients with de novo renal transplant.

Renal function will be accurately evaluated by measuring the clearance of iohexol.

The protocol will also evaluate the efficacy and safety in a short term of these two different immunosuppressive regimens.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged between 18 and 70.
* Patient receiving a first or second kidney transplant from a deceased donor, living related or unrelated.
* Patient with a maximum PRA <20%.
* Patient wishing and being able to participate fully to the study, and having given a written consent.
* Patient covered by a social insurance or beneficiary of such a regime.
* Women of childbearing age must use a recognized method of contraception throughout the study period and continue for 8 weeks after discontinuation of study treatment.

Exclusion Criteria:

* Patient receiving a kidney from a heart attack donor , or an ABO incompatible donor or a donor with a positive T-cross match.
* Patient with a maximum PRA> 20% twice.
* Cold ischemic time > 36 hours.
* Patients with thrombocytopenia (<75000/mm3), neutropenia (<1 500 / mm3), leukopenia (<2 500 / mm3) or a hemoglobin concentration <8 g / dl, at inclusion visit.
* Patient with severe hyperlipidemia: total cholesterol ≥ 9 mmol / l (≥ 3.50 g / l) and / or triglycerides ≥ 8.5 mmol/l (≥ 7.5 g / l) despite appropriate lipid-lowering therapy.
* Patient with known HIV positive status, know active hepatitis B or C. Recipients of an organ from a donor with positive HIV status, hepatitis B or hepatitis C are excluded.
* Patient with severe systemic infections requiring continued therapy.
* Treatment with an experimental drug within 4 weeks before the first dose of study treatment.
* Patient for whom the initial disease or other pathology requires a long-term corticosteroid treatment.
* Patient with a history of hypersensitivity or known contra-indications for macrolide or inhibitors of mTORs drugs; drugs similar to Myfortic ® (ERL080) or other components of the formulation such as lactose, or cyclosporine, or prednisone (Cortancyl ®), or Thymoglobuline ® or Iohexol.
* Patient with a malignant disease or a history of malignancy over the past 5 years except squamous-cell or basal cell carcinoma wich was excised.
* Medical condition or surgical procedure, except transplantation, which could exclude the patient in the opinion of the investigator.
* Patient with symptoms of mental or significant somatic illness. Disability to cooperate or communicate with the investigator.
* Pregnant, sucking or of childbearing age and refusing or being unable to use a recognized contraceptive method.
* Patient under guardianship, or any patient protected by law.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Evolution of glomerular filtration rate measured by clearance of iohexol | one year

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nephrology department, Hospital University of Amiens, Amiens
  - Nephrology Department, University Hospital of Montpellier, Montpellier